CLINICAL TRIAL: NCT00906412
Title: VIM DBS and Working Memory
Brief Title: Ventrointermediate Nucleus (VIM DBS) and Working Memory
Acronym: WMVIM
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0732
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Essential Tremor
Keywords: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ET Group: Total of 25 participants with ET
- Controls: 25 controls without ET

SUMMARY:
This is part of a larger study for which participants have already completed memory and thinking tests. In this study, investigators are trying to learn how deep-brain stimulation affects memory skills in essential tremor (ET) patients. We are especially trying to figure out how stimulation on each side of the brain may affect working memory.

ELIGIBILITY:
Inclusion Criteria:

ET PATIENTS:

* Clinical diagnosis of essential tremor affecting the upper extremities.
* Previous unilateral or bilateral DBS of the VIM
* Ages 40 -70
* A useable pre-surgical MR scan

CONTROLS:

* Spouse or acquaintance of enrolled patient participant
* Ages 40 - 70

Exclusion Criteria:

ET PATIENTS:

* Clinical evidence of other neurological conditions
* Significant psychiatric condition

CONTROLS:

* Clinical evidence of other neurological conditions
* Significant psychiatric condition

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Washington University School of Medicine Movement Disorder Clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2013-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hershey Tamara, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and consent to share data was not obtained.